CLINICAL TRIAL: NCT00328640
Title: Secondary Prevention After Ischemic Stroke: A Trial of an Evidence-Based System-Wide Intervention
Brief Title: Quality Improvement in Stroke Prevention (QUISP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: MM 0620 0404
Record Dates: First submitted 2006-05-18; First posted 2006-05-22 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Ischemic Stroke
Keywords: CVA; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Optimal treatment

SUMMARY:
Is a secondary prevention intervention, focused on implementation of standardized pre-printed discharge orders for hospitalists, effective at increasing utilization of the following evidence-based treatments 6 months after discharge for ischemic stroke:

1. Treatment with statins,
2. Control of hypertension, and
3. Anticoagulation in patients with atrial fibrillation.

DETAILED DESCRIPTION:
There are several proven strategies for prevention of recurrent ischemic stroke, including use of statins, treatment of hypertension, and anticoagulation in patients with atrial fibrillation. Preliminary analyses suggest that only 9-15% of Kaiser Permanente Northern California's ischemic stroke patients receive optimal care for secondary prevention of stroke. The purpose of this study is to determine whether or not a quality improvement (QI) intervention can improve the care received by stroke patients. This project consists of a randomized trial of standardized stroke discharge order forms to improve adherence with best practices in secondary stroke prevention. The primary research question is: Is a secondary prevention intervention, focused on implementation of standardized pre-printed discharge orders for hospitalists, effective at increasing utilization of the following evidence-based treatments 6 months after discharge for ischemic stroke: (1) treatment with statins, (2) control of hypertension, and (3) anticoagulation in patients with atrial fibrillation.

The primary outcome will be the proportion of patients receiving optimal treatment, as defined by these three goals. The impact of the intervention will be measures as a change after-to-before at intervention hospitals compared to non-intervention (control) hospitals, with the institution as the unit of analysis. Secondary analyses will evaluate the impact of the intervention on each of these components and on 6-month and 1-year rates of mortality, readmission for stroke, and costs of care after discharge.

ELIGIBILITY:
Inclusion Criteria:

Ischemic stroke Kaiser-Permanente Health Plan Member with Pharmacy Benefit Discharged alive to home

Exclusion Criteria:

tpA patients Hemorrhagic stroke TIA Significant comorbidities

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2005-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Medication utilization
Best Practices
Recurrent stroke

SECONDARY OUTCOMES:
Mortality
Morbidity
Cost
Hospital readmission

CONTACTS AND LOCATIONS:
Overall Officials: David M Grosvenor, MPH, Study Director — University of California, San Francisco; S C Johnston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kaiser-Permanente Division of Research, Oakland, California, United States

REFERENCES:
- [Derived] Johnston SC, Sidney S, Hills NK, Grosvenor D, Klingman JG, Bernstein A, Levin E. Standardized discharge orders after stroke: results of the quality improvement in stroke prevention (QUISP) cluster randomized trial. Ann Neurol. 2010 May;67(5):579-89. doi: 10.1002/ana.22019. PMID 20437555